CLINICAL TRIAL: NCT07379476
Title: ATOM2: A Randomized Phase II Trial on Ablative Therapy to Oligoresidual Metastasis in EGFR Mutated Non-small Cell Lung Cancer After Osimertinib Treatment
Brief Title: Local Ablative Therapy to Oligoresidual Metastasis in EGFR Mutated Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Molly SC Li, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUN126
Record Dates: First submitted 2025-12-17; First posted 2026-01-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy arm (Experimental): * Continue osimertinib as per standard of care (40mg or 80mg daily).
  * Undergo radiotherapy to 1-3 disease sites as determined by the investigator.
  Interventions: Radiation: Local ablative therapy
- Control arm (Active Comparator): Continue osimertinib as per standard of care (40mg or 80mg daily)
  Interventions: Drug: Osimertinib alone

INTERVENTIONS:
Radiation: Local ablative therapy — Local ablative therapy (LAT) will be given in the form of stereotactic body radiotherapy (SBRT) or hypofractionated radiotherapy. LAT should be started within 90 days from the screening PET-CT scan.
  Arms: Radiotherapy arm
Drug: Osimertinib alone — Continue osimertinib as per standard of care (40mg or 80mg daily)
  Arms: Control arm

SUMMARY:
This is an open-label, multicentre, randomized phase II clinical trial. Patients with stage IV (AJCC 9th edition) non-small cell lung cancer (NSCLC) harboring EGFR exon 19 deletion or exon 21 L858R mutation, who had less than or equal to 3 active oligoresidual cancer sites amenable to local ablative therapy (LAT) (as determined by physician) after 3-6 months of firstline osimertinib treatment, are eligible. Subjects will be randomized 1:1 to osimertinib with or without LAT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and able to understand and give written informed consent
* Pathologically proven non-small cell lung cancer
* Positive for EGFR exon 19 deletion or EGFR exon 21 L858R mutation (either by tissue or plasma testing)
* Stage IV disease
* Receive first line osimertinib monotherapy for stage IV disease
* Undergo a PET-CT scan after 12-24 weeks of initiation of osimertinib treatment, with no evidence of disease progression, and less than or equal to 3 active disease sites (including primary tumour) amenable to local ablative therapy, as determined by investigator
* At least one brain imaging (CT Brain or MRI Brain with contrast, preferably MRI Brain), either at time of diagnosis or while on osimertinib treatment but before randomization, to document CNS status for stratification. Patients with asymptomatic CNS metastases are eligible. For patients with brain metastases diagnosed at baseline, follow up brain imaging is recommended before randomization.
* Patients with history of palliative radiotherapy are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate haematological values: haemoglobin ≥9.0g/dL, absolute neutreophil count ≥1.0 x 109/L, platelet count ≥100 x 109/L
* Adequate hepatic function: bilirubin ≤1.5 x ULN, AST/ALT ≤2.5 x ULN
* Adequate renal function: creatinine clearance ≥30ml/min, according to the formula of Cockcroft-Gault equation
* Willing and able to comply with the requirements and restrictions in this protocol

Exclusion Criteria:

* Previous or concomitant malignancy within 5 years prior registration with the exception of adequately treated localized non-melanoma skin cancer or cervical cancer in situ.
* Mixed SCLC and NSCLC histology
* Positive pregnancy test
* Contraindication to radiotherapy
* Any serious underlying medical, psychiatric, psychological, familial condition that in the judgement of the investigator, that may interfere with planned staging, treatment and follow up, affect patient compliance, or place the patient at high risk from treatment related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-02-11 (Actual); Primary Completion 2029-03-03 (Estimated); Study Completion 2030-03-03 (Estimated)

PRIMARY OUTCOMES:
18 month progression-free survival rate (PFS) in per-protocol population as determined by investigator. | up to 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
Safety and tolerability reflected by number of participants with treatment related adverse events as assessed by CTCAE v5.0, number of participants with SAE | 2 years
Time to treatment failure (TTF), defined as the time period between osimertinib initiation and cessation or death | 2 years
Site of tumour progression at disease progression | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No